CLINICAL TRIAL: NCT07155642
Title: Effects of Yoga and Conventional Physiotherapy Programs on Fatigue, Balance, Walking and Quality of Life in Multiple Sclerosis Patients.
Brief Title: Yoga in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Nursel Oziri, PhD, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRU-FTR-NO-02
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; yoga; fatigue; balance; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga (Experimental): Participants in the yoga group received a total of 8 weeks of intervention, conducted 3 days a week, for 60 minutes per day. The program components were:
  * 8 minutes of meditation practice.
  * 40 minutes of Yin and Yang yoga postures. (It's highly recommended to briefly explain what "Yin and Yang yoga postures" specifically entail in the full paper's methodology section, e.g., "Yin yoga focuses on holding passive poses for longer durations to target deep connective tissues, while Yang yoga incorporates more active, flowing sequences to build strength and flexibility.")
  * 2 minutes of breathing exercises (pranayama).
  * 10 minutes of deep relaxation (savasana).
  Interventions: Other: yoga
- Conventional Physiotherapy (Active Comparator): Participants in the conventional physiotherapy group also underwent an 8-week program, 3 days a week, for 60 minutes per day. This program included:
  * Aerobic exercises.
  * Stretching exercises.
  * Strengthening exercises.
  * Spinal stabilization exercises.
  * Balance exercises.
  Interventions: Other: conventional physiotheraphy

INTERVENTIONS:
Other: yoga — Participants in the yoga group received a total of 8 weeks of intervention, conducted 3 days a week, for 60 minutes per day. The program components were: • 8 minutes of meditation practice. • 40 minutes of Yin and Yang yoga postures. (It's highly recommended to briefly explain what "Yin and Yang yoga postures" specifically entail in the full paper's methodology section, e.g., "Yin yoga focuses on holding passive poses for longer durations to target deep connective tissues, while Yang yoga incorporates more active, flowing sequences to build strength and flexibility.") • 2 minutes of breathing exercises (pranayama). • 10 minutes of deep relaxation (savasana).
  Arms: yoga
Other: conventional physiotheraphy — Participants in the conventional physiotherapy group also underwent an 8-week program, 3 days a week, for 60 minutes per day. This program included:
  * Aerobic exercises.
  * Stretching exercises.
  * Strengthening exercises.
  * Spinal stabilization exercises.
  * Balance exercises.
  Arms: Conventional Physiotherapy

SUMMARY:
Objective

The objective of this study will be to compare the effects of an eight-week Yin-based yoga program and conventional physiotherapy on fatigue, balance, gait, and quality of life in individuals with Multiple Sclerosis (MS).

Methods

Twenty patients with MS will be randomly assigned to either a yoga group (n = 10) or a physiotherapy group (n = 10). Both groups will participate in supervised sessions lasting 60 minutes per day, three days per week, over an eight-week period.

The yoga intervention will be Yin-based, incorporating centering, yoga postures, breathing exercises, and relaxation.

The physiotherapy program will consist of aerobic training, strengthening and spinal stabilization exercises, balance and coordination activities, and stretching.

Outcome measures will include the Fatigue Severity Scale (FSS) for fatigue, the Berg Balance Scale (BBS) for balance, the 12-item Multiple Sclerosis Walking Scale (MSWS-12) for gait, and the Multiple Sclerosis Quality of Life Questionnaire (MSQOL-54) for physical and mental health-related quality of life.

DETAILED DESCRIPTION:
Intervention Protocol Yoga Program

The yoga intervention will be implemented in small groups of up to five participants, three times per week for a duration of eight weeks. Sessions will be led by a physiotherapist experienced in working with multiple sclerosis (MS) patients and certified in yoga practice. Each session will last 60 minutes and will consist of four structured components:

Centering/Meditation (5-10 minutes):

Participants will perform breath-focused meditation in a comfortable seated position, using cushions if required. The duration will begin at 5 minutes during the first week and will gradually increase to 8-10 minutes by the third week. Participants will be instructed to count their breaths up to ten, restarting from one if their focus drifts.

Yin and Yang Yoga Poses (40 minutes):

This segment will combine Yin poses (passive, long-held postures targeting connective tissues) and Yang poses (active, dynamic postures).

Yin poses: Held for 2-3 minutes.

Yang poses: Will include Bridge, Plank, Low Lunge, Crescent Lunge, Cat-Cow, Downward-Facing Dog, and Chair Pose. These will be held for 10-30 seconds and repeated at least three times.

Rest periods of 30-60 seconds in Child's Pose will be incorporated between sequences. Postures will be adapted according to individual needs and physical capacities, applying the "soft edge" principle to avoid discomfort. Props such as blocks will be used as needed. Both verbal and tactile corrections will be provided.

Breathing Exercises (Pranayama) (1-2 minutes):

Alternating Nostril Breathing (Nadi Shodhana) will be practiced to balance the effects of Yin and Yang postures.

Deep Relaxation (Savasana) (10 minutes):

Sessions will conclude with Savasana, in which participants will lie supine for 10 minutes with arms relaxed at the sides and palms facing upward, maintaining complete stillness and relaxation.

During yoga sessions, the room temperature will be maintained at 23-26°C, and soft, relaxing music will be played.

Physiotherapy Program

Participants assigned to the physiotherapy group will receive individualized, exercise-based interventions designed to address aerobic capacity, muscle strength, spinal stabilization, balance, coordination, and flexibility. The intervention will be structured as follows:

Aerobic Exercise (10 minutes):

Horizontal cycling will be performed at a submaximal heart rate (60-80% of average). Room temperature will be kept at 20-22°C to prevent overheating.

Strengthening and Spinal Stabilization Exercises (20 minutes):

Exercises will target large muscle groups of the lower extremities (dorsiflexors, knee and hip extensors), the spine, and the shoulder girdle. Training will begin with 8-10 repetitions at 60-80% of one repetition maximum, progressing to two sets by week 2 and 15 repetitions by week 4. Resistance will be increased by 2-5% every three weeks. Rest intervals of 2-4 minutes will be allowed between exercises. Tactile feedback and instruction will be provided to ensure correct spinal stabilization techniques.

Balance and Coordination Exercises (20 minutes):

Training will progress from static to dynamic balance and will include dual-task activities. Difficulty will be gradually increased by performing tasks with eyes open and closed, shifting the center of gravity, and utilizing various balance-training materials. External support will be progressively reduced to encourage independence while maintaining motivation.

Stretching Exercises (10 minutes):

The final component of each session will involve active stretching of the hamstrings, hip flexors, adductors, quadriceps, and plantar flexors. Each stretch will be held for 20-60 seconds within the comfortable range of motion, ensuring that no pain is experienced. Straps will be provided as supportive aids when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age.
* Voluntarily giving informed consent to participate in the study.
* Having either Relapsing-Remitting MS (RRMS) or Secondary Progressive MS (SPMS) type.
* An Expanded Disability Status Scale (EDSS) score of 5.5 or below.
* No MS exacerbation within the last 4 weeks.
* Possessing the willingness, ability, and cognitive intactness to participate in the interventions.

Exclusion Criteria:

* Using medication specifically for fatigue.
* Presence of major sleep disorders, clinical depression, hypothyroidism, or B12 deficiency.
* Severe balance problems (e.g., Central Vestibular Disorders (CVO), peripheral neuropathy, Meniere's disease, vertigo).
* Having received corticosteroid treatment within the last 4 weeks.
* Pregnancy.
* Serious cardiovascular disease, hypertension, or orthopedic limitations.
* Presence of Carpal Tunnel Syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
MS Walking Scale (MSWS-12) | 3 months
  The MSWS-12 is a 12-item self-reported questionnaire that assesses the impact of MS on walking ability over the past two weeks. Items are rated on a 5-point scale (1: almost never, 5: extremely). Higher scores indicate greater perceived walking limitations or difficulties
MS Quality of Life-54 (MSQOL-54) | 3 months
  The MSQOL-54 is a disease-specific quality of life questionnaire for MS patients. It comprises 31 questions divided into three sub-dimensions: psychological, physical, and psychosocial quality of life. Lower scores indicate a higher quality of life

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | 3 months
  The FSS is a 9-item scale used to quantify fatigue. Each item is scored from 1 (strongly disagree) to 7 (strongly agree), and the total score is calculated as the average of the nine items. A score of 4 or higher indicates pathological fatigue. Lower scores indicate less severe fatigue
Berg Balance Scale (BBS) | 3 months
  The BBS is a 14-item objective measure used to assess balance abilities. Each item is scored from 0 (unable to perform) to 4 (independently performs), yielding a maximum total score of 56. Scores between 0-20 indicate a high fall risk, 21-40 a moderate fall risk, and 41-56 a low fall risk. The test utilizes common items such as steps, a ruler, a stopwatch, and a chair to evaluate postural control and fall risk

CONTACTS AND LOCATIONS:
Locations (1):
- Öziri, Ataşehir, Istanbul, Turkey (Türkiye)